CLINICAL TRIAL: NCT04339218
Title: Cryoablation in Combination (or Not) With Pembrolizumab and Pemetrexed-carboplatin in First-line Treatment for Patients With Metastatic Lung Adenocarcinoma: A Randomized Phase III Study
Brief Title: Cryoablation in Combination (or Not) With Pembrolizumab and Pemetrexed-carboplatin in 1st-line Treatment for Patients With Metastatic Lung Adenocarcinoma
Acronym: CRYOMUNE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2019-05; 2019-A02477-50 (Other: ANSM ID-RCB number)
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Lung Adenocarcinoma; Cryotherapy Effect
Keywords: Lung adenocarcinoma, immunotherapy, cryoablation
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Cryosurgery; pembrolizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Cryoablation+pembrolizumab-pemetrexed-carboplatin (Experimental): Cryoablation of one visceral lesion or bone metastasis excluding liver and sclerotic bone metastases combined with pembrolizumab and pemetrexed-carboplatin prescribed as per market authorization.
  Interventions: Device: Cryoablation; Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin
- Arm pembrolizumab-pemetrexed-carboplatin (Active Comparator): Combination of Pembrolizumab and pemetrexed-carboplatin prescribed as per market authorization.
  Interventions: Drug: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Device: Cryoablation — Cryoablation will be performed by a specialized radiologist, percutaneously, ie "through the skin". The operation is performed under general anesthesia, under the guidance of the scanner. The images from the scanner make it possible to precisely insert and place a needle at the level of the tumor to be treated. Intense cold will be produced by the needle and will destroy the cancer cells by freezing (temperatures of -40 °C). Freezing is localized to the tumor, the rest of the organ will not suffer from the cold.
  The aftermath of the intervention causes only minimal pain and in most cases does not require pain treatment. As the operation is minimally traumatic, the risk of complications is low. Hospitalization is around twenty-four hours and usual or professional activities can be resumed very quickly.
  Arms: Arm Cryoablation+pembrolizumab-pemetrexed-carboplatin
Drug: Pembrolizumab — Pembrolizumab will be prescribed and administered at the dose recommended by market authorization.
Drug: Pemetrexed — Pemetrexed will be prescribed and administered at the dose recommended by market authorization.
Drug: Carboplatin — Carboplatin will be prescribed and administered at the dose recommended by market authorization.

SUMMARY:
This study aims to compare the one-year survival benefit of the association of cryoablation-pembrolizumab-pemetrexed-carboplatin versus pembrolizumab-pemetrexed-carboplatin in metastatic lung adenocarcinoma patients.

This is a multicenter, prospective, open-labeled, 2-arm comparative randomized (1:1) phase III trial.

Patients will be randomized with a 1:1 ratio into:

* Arm A (experimental arm): cryoablation of one visceral lesion or bone metastasis excluding liver and sclerotic bone metastases combined with pembrolizumab and pemetrexed-carboplatin prescribed as per market authorization.
* Arm B (standard arm): pembrolizumab and pemetrexed-carboplatin prescribed as per market authorization.

Pembrolizumab and pemetrexed-carboplatin will be prescribed and administered at the dose recommended by market authorization.

Cryoablation treatment should be performed within 6 weeks after the first administration of pembrolizumab. No treatment switching permitted.

DETAILED DESCRIPTION:
Upon signature of the informed consent and verification of the screening results, eligible participants will be randomized between two therapeutic strategies:

* Arm A (experimental arm): cryoablation of visceral lesion or bone metastasis excluding liver and sclerotic bone metastases combined with pembrolizumab and pemetrexed-carboplatin prescribed as per market authorization.
* Arm B (standard arm): pembrolizumab and pemetrexed-carboplatin prescribed as per market authorization.

Pembrolizumab treatment should begin no later than 7 days after randomization. The cryoablation treatment should be performed within 6 weeks after the first administration of pembrolizumab.

RECIST v1.1 tumour assessment:Tumour response will be defined and assessed as per the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

* A comprehensive workup will be performed at baseline and every 9 weeks.
* The same method will be used to evaluate each identified lesion both at baseline and throughout the study.
* Treatment will be administered as long as no disease progression or unacceptable toxicity is found, or as long as no other reasons for treatment discontinuation are met.
* Assessment of efficacy will be essentially based on a set of measurable lesions identified at baseline as target lesions and followed until disease progression and following the RECIST v1.1 criteria.
* Confirmation of response at least 4 weeks later is not required in this randomized study where response is not the primary endpoint.

SAFETY :Patients will be evaluable for safety if they have received at least one treatment administration. Safety profile will be continuously followed during treatment up to 90 days after the last immunotherapy treatment administration or until the start of a new antitumor therapy or until 12 months of treatment, whichever occurs first.

STUDY PROCEDURES :

Blood sample will be collected at baseline (Day 1: before treatment initiation), Day 1 cycle 2 (Day 21 +/- 3 days), Day 1 cycle 3 (Day 42 +/- 3 days) and progression.

Patients will be asked to provide samples of biopsy tissue at screening (prior to anticancer agent with immunomodulatory activity treatment initiation), during treatment (day 42 +/- 3 days) and at disease progression as follows. Tumor biopsy at inclusion is optional if materiel archived fixed in formalin and embedded in paraffin of diagnostic biopsy is available.

All randomized patients will be followed up until death or the end of the follow-up period, defined as 36 months after randomization, whichever occurs first. For all patients, treatments regimen, tumor response during and/or after treatment, survival follow-up will be collected on study database:

* Every 3 months until loco-regional relapse or metastasis evidence, death or until the date of study termination, whichever occurs first,
* Every 6 months after loco-regional relapse or metastasis evidence, until death or until the date of study termination, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-small lung adenocarcinoma.
2. Metastatic disease.
3. Treatment with pembrolizumab in combination with pemetrexed-carboplatin as per market authorization.
4. At least two target lesions (RECIST1.1), measurable with CT or MRI :

   1. One target lesion that is amenable for accurate repeated measurements,
   2. One target lesion (15-40 mm) that is amenable for cryoablation treatment including lung, kidney, adrenal, soft tissue and lytic bone lesions. Liver and sclerotic bone lesions are not allowed to be treated by cryoablation.
5. Age ≥ 18.
6. Performance status ≤ 2.
7. Women of childbearing potential must have a negative serum pregnancy test prior to registration.
8. Recovery to grade ≤ 1 from any adverse event derived from previous treatment (excluding alopecia)
9. Patients with a social security in compliance with the French law (Loi Jardé).
10. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
11. Voluntarily signed and dated written informed consents prior to any study specific procedure.

Exclusion Criteria:

1. Squamous cell tumors and other than adenocarcinoma.
2. Prior systemic treatment for advanced non-small cell lung cancer (except adjuvant therapy after complete resection).
3. Current or prior use of immunosuppressive medication including any use of oral glucocorticoids, within 21 days before the first dose of pembrolizumab.
4. Known contra-indication and/or hypersensitivity to PD1/PD-L1 antagonist and/or cytotoxic therapy.
5. Known contra-indication to cryoablation.
6. Abnormal coagulation contraindicating biopsy.
7. Prior or concurrent malignant disease diagnosed or treated in the last 2 years except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma or incidentally discovered good prognosis prostate cancer (T stage < pT3 and Gleason ≤ 7).
8. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
9. Subjects who participated in an investigational drug or device study within 28 days prior to study entry.
10. Known infection with HIV, hepatitis B, or hepatitis C.
11. Females who are pregnant or breast-feeding.
12. Men or women refusing contraception.
13. Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
14. Previous enrolment in the present study.
15. Individuals deprived of liberty or placed under legal guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2028-08-27 (Estimated)

PRIMARY OUTCOMES:
1-year overall survival rate | 1 year
  Overall survival (OS) is defined as the time interval between the date of randomization and the date of death (from any cause). Patients alive will be censored at the date of last follow-up or last patient contact. One-year OS rates will be compared between arms.

SECONDARY OUTCOMES:
Overall response rate within 6 months as per RECIST v1.1 | throughout the treatment period, an expected average of 6 months
  Overall response rate (ORR) is defined as the rate of patients with complete or partial response (CR, PR) as per RECIST v1.1. According to RECIST v1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.; Overall Response (OR) = CR + PR.
Overall response rate at 6 months as per RECIST v1.1 | 6 months
  Overall response rate (ORR) is defined as the rate of patients with complete or partial response (CR, PR) as per RECIST v1.1. According to RECIST v1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.; Overall Response (OR) = CR + PR.
Overall response rate as per RECIST v1.1 | throughout the treatment period, an expected average of 1 year
  Overall response rate (ORR) is defined as the rate of patients with complete or partial response (CR, PR) as per RECIST v1.1. ORR will be assessed across all time points, once all the data for the patient is known. According to RECIST v1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.; Overall Response (OR) = CR + PR.
Duration of overall response | throughout the treatment period, an expected average of 1 year
  The duration of overall response (DoR) is defined as the time from documentation of tumour response (Complete or partial responses whichever is first recorded) to disease progression, according to RECIST v1.1. Kaplan-Meier Method will be used to estimate DoR.
Best overall response rate as per RECIST v1.1 | throughout the treatment period, an expected average of 1 year
  Best overall response rate (BoR) is defined as rate of patients with the best response across all time points (RECIST v1.1). The best overall response will be determined once all the data for the patient is known.
2-year overall survival rate | 2 years
  Overall survival (OS) is defined as the time interval between the date of randomization and the date of death (from any cause). 2-year OS rates will be compared between arms.
1-year progression-free survival rate | 1 year
  Progression-free survival (PFS) is defined as the time interval between the date of randomization and the date of progression (RECIST v1.1) or death (from any cause), whichever occurs first.The analysis of PFS will be based on the censoring process following FDA guidelines. Progression is defined using RECIST v1.1, as a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), or a unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.1-year PFS rates will be compared between arms.
2-year progression-free survival rate | 2 years
  Progression-free survival (PFS) is defined as the time interval between the date of randomization and the date of progression (RECIST v1.1) or death (from any cause), whichever occurs first.The analysis of PFS will be based on the censoring process following FDA guidelines. Progression is defined using RECIST v1.1, as a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study), or a unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.2-year PFS rates will be compared between arms.
Mean scores of each dimension of QLQ-C30 from EORTC quality of life group | at baseline, 3, 6, 9, 12 and 24 months
  Health-related quality of life (HRQoL) will be assessed through EORTC QLQ-C30 (Aaronson et al. J Natl Cancer Inst 1993).The QLQ-C30 is a questionnaire developed to assess the quality of life of cancer patients. The questionnaire includes one global health status/QoL scale, five functional scales and three symptom scale. Each scale is scored from 0 to 100. A high score on a scale indicate a good outcome for the dimension of QoL.
Time to health-related quality of life score definitive deterioration (targeted dimension of EORTC QLQC30 : global health) | at baseline, 3, 6, 9, 12 and 24 months
  Time until definitive deterioration (TUDD) of HRQoL is defined as the time from the date of randomization to a first deterioration of at least 10 points of HRQoL as compared to the baseline score (Bonnetain et al. Eur J Cancer 2010).
Number of patient receiving a post-progression treatment | an average of 6 months
  Post-progression treatment is defined as the treatment (systemic/local) given after the first progression under cryoablation+pembrolizumab and pemetrexed-carboplatin or pembrolizumab and pemetrexed-carboplatin.
Overall response rate as per iRECIST | throughout the treatment period, an expected average of 6 months
  Overall response rate (ORR) is defined as the rate of patients with immune complete or partial responses (iCR, iPR) as per iRECIST (Seymour et al. 2017). iCR and iPR can be assigned after iUPD (immune unconfirmed progressive disease) has been documented.
Duration of immune overall response | throughout the treatment period, an expected average of 1 year
  Duration of i-response (iDoR) is defined as the time from the date of the first response iCR/iPR (whichever is first recorded) to the date of PD (iUPD confirmed as iCPD). iDOR is only defined for subjects who have best overall response of iCR or iPR.
1-year immune-progression-free survival rate | 1 year
  Immune-progression-free survival (iPFS) is defined as the time interval between the date of randomization and the date of progression (iRECIST) or death (from any cause), whichever occurs first. The event date to be used for calculation of progression-free survival (iPFS) should be the first date at which progression criteria are met (ie, the date of iUPD) provided that iCPD is confirmed at the next assessment. 1-year iPFS rates will be compared between arms.
2-year immune-progression-free survival rate | 2 year
  Immune-progression-free survival (iPFS) is defined as the time interval between the date of randomization and the date of progression (iRECIST) or death (from any cause), whichever occurs first. The event date to be used for calculation of progression-free survival (iPFS) should be the first date at which progression criteria are met (ie, the date of iUPD) provided that iCPD is confirmed at the next assessment. 2-year iPFS rates will be compared between arms.
Best overall response rate as per iRECIST | throughout the treatment period, an expected average of 1 year
  Best overall response rate (iBoR) is defined, according to iRECIST, as the rate of patients with the best timepoint response recorded from the start of the study treatment until the end of treatment, taking into account any requirement for confirmation.
Number of immune-related SAEs (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Serious Adverse events (SAEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of immune-related AEs (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Adverse events (AEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of chemotherapy-related SAEs (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Serious Adverse events (SAEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of chemotherapy-related AEs (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Adverse events (AEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of cryoablation-related SAEs (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Serious Adverse events (SAEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of cryoablation-related AEs (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Adverse events (AEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of SAEs related to study procedures (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Serious Adverse events (SAEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of AEs related to study procedures (CTCAE NCI V5) | throughout the treatment period, an expected average of 1 year
  Adverse events (AEs) will be coded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE) NCI v5.
Number of hospitalisations in experimental arm only | within 6 weeks + 30 days after first pembrolizumab administration
  counts of hospitalisations within 30 days after the cryoablation will be summarized by treatment strategy.
Percentage of patients that worsen their ECOG score of 1 or more point | at follow-up visits post randomization (an average of 2 years)
  Percentage of patients that worsen their ECOG score of 1 or more point at follow-up visits post randomization will be summarized by treatment strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean PALUSSIERE, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié, Bordeaux, Gironde, France